CLINICAL TRIAL: NCT03923569
Title: Epileptiform Activity During REM Sleep in Alzheimer's Disease
Acronym: EREMAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre de Recherches sur la Cognition Animale (CRCA - UMR5169 CNRS/UPS) (Unknown); Centre de Recherche Cerveau & Cognition (CerCo - UMR5549 CNRS/UPS) (Unknown); Toulouse NeuroImaging Center (ToNIC - UMR 1214 Inserm/UPS) (Unknown); Fondation Plan Alzheimer (Other); IHNPS/FHU HoPeS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/18/0265; 2018-A02229-46 (Other: ID RCB)
Record Dates: First submitted 2019-03-29; First posted 2019-04-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer's disease; Rapid eye movement (REM) sleep; Memory consolidation; Epilepsy; MRI
MeSH Terms: conditions — Alzheimer Disease; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 2 compared groups (Alzheimer's Disease patients vs controls)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer's Disease patients group (Other): This group contains the 31 (anticipated) participants with a diagnosis of Alzheimer's disease
  Interventions: Diagnostic Test: Overnight polysomnography; Diagnostic Test: blood sample; Diagnostic Test: high-resolution MRI scan; Behavioral: neuropsychological evaluation
- Healthy control group (Other): This group contains the 31 (anticipated) age and sex -matched healthy controls
  Interventions: Diagnostic Test: Overnight polysomnography; Diagnostic Test: high-resolution MRI scan; Behavioral: neuropsychological evaluation

INTERVENTIONS:
Diagnostic Test: Overnight polysomnography — Overnight polysomnography with evaluation of each form of epileptiform activity during each vigilance state and memory scores at the overnight retention test
Diagnostic Test: blood sample — blood sample for genetic testing of the Apolipoprotein E
  Arms: Alzheimer's Disease patients group
Diagnostic Test: high-resolution MRI scan — Evaluation of anomalies in brain structure and functional resting state connectivity
Behavioral: neuropsychological evaluation — neuropsychological evaluation including episodic memory tests before an overnight polysomnography

SUMMARY:
Recent clinical data showed that patients with Alzheimer Disease (AD) might present epilepsy at early stages of the disease (Cretin et al., 2016, Vossel et al., 2016). In mice models of Alzheimer disease, preclinical researchers observed an increase of epileptic events during Rapid Eye Movement (REM) sleep, which is very unusual. This study aims at testing if patients with AD present an exacerbation of epileptic events during REM sleep, which could constitute an early biomarker of the disease. Investigators will evaluate the incidence of epilepsy during each sleep stage in 40 patients with early or moderate forms of AD and in 40 healthy subjects. Investigators will also look for a link between epilepsy during sleep in AD participants and memory performances, brain damage (by using MRI scans) and in the case of patients, the phenotype of the Apolipoprotein E(ApoE) gene.

DETAILED DESCRIPTION:
Preclinical researchers discovered that the Tg2576 mouse model of Alzheimer Disease (AD) presents epileptiform activity specifically during sleep, with a prominent increase during REM-sleep. This phenotype is specific to AD mice since REM-sleep usually prevents seizures and epileptiform activity in animal models of epilepsy. Preclinical research also evidenced that this epileptic phenotype occurs at very early age in Tg2576 mice, far before the onset of cognitive impairments. Thus, it was hypothesized that patients with AD might present subclinical epileptiform events during sleep with a potential worsening during REM-sleep. If so, it could be used as a specific and early biomarker of AD. Since sleep is involved in memory consolidation processes, preclinical researchers also hypothesized that epileptiform events during sleep might participate to cognitive dysfunction in AD patients.

In order to test this hypothesis, a monocentric clinical study with a protocol consisting of three visits was designed aiming at evaluating seizures and subclinical epileptiform activity - and their consequences on memory - during sleep in 31 patients at early to moderate stages of AD and 31 matched healthy participants. During the first visit, a blood sample is collected of each patient for genetic testing of the ApoE gene before they undergo a high-resolution MRI scan. During the second visit (in the 60 days following the first one) participants first undergo a neuropsychological evaluation including visual, verbal and episodic memory tests before an overnight polysomnography. Following the overnight polysomnography, all subjects (patients and healthy participants) will be tested for the memories acquired the day before in order to evaluate sleep related memory consolidation. During the last visit, participants will fill out questionnaires aiming at evaluating pre-diagnostic lifestyle and they (and one family member if possible) will be interviewed about the presence of symptoms that might indicate an underlying epileptic syndrome for the participant. Healthy subjects will undergo the same procedures except for the blood test from which they will be exempted.

This should allow to evidence sleep related epileptic events, to precise their incidence in AD patients as well as in healthy participants, and to correlate these events to anomalies in brain structure and functional resting state connectivity (MRI) and/or sleep disturbances and/or cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* age from 50 to 90 years old
* affiliated to the French health care system

For AD patients:

* meeting International Working Group (IWG)-2 criteria for diagnosis
* Mini-Mental State Examination (MMSE) ≥18 (Greco version)

For healthy volunteers:

* MMSE>25
* Dubois 5 words test ≥ 9

Exclusion Criteria:

For all participants:

* Pregnancy
* people not able to give consent
* contraindication for MRI (metallic body parts, claustrophobia),
* aphasia, apraxia or agnosia
* neurological (other than AD) or any other serious disease (cancer, addiction, systemic disease)
* non treated sleep apnea
* major depression or anxiety for more than 3 months (Beck>10) or psychiatric disease
* documented epilepsy
* use of neuroleptics (more than one dose per day)
* use of antiepileptics
* use of benzodiazepines at a dose superior or equal to two intakes per day
* use of antidepressants
* restless leg syndrome treated by dopaminergic agonists.

For AD patients:

* other causes of dementia
* non-degenerative neurological lesions
* white matter hypersignals
* acute cognitive deficits

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Epileptiform activity during REM sleep | Day 2
  the proportion of participants from each group exhibiting a significant epileptiform activity (seizures and/or interictal spikes) during REM sleep.
  . Epileptiform activity will be defined as either at least one spike, or at least 4 paroxysmal activities.

SECONDARY OUTCOMES:
Number of epileptiform activity according to sleep-wake cycle | Day 2
  Number of epileptiform activity according to sleep-wake cycle in each group
Frequency of epileptiform activity according to sleep-wake cycle | Day 2
  Frequency of epileptiform activity according to sleep-wake cycle in each group
lateralization of epileptiform activity according to sleep-wake cycle | Day 2
  lateralization of epileptiform activity according to sleep-wake cycle in each group
localization of epileptiform activity according to sleep-wake cycle | Day 2
  localization of epileptiform activity according to sleep-wake cycle in each group
Comparison of sleep characterization between the two groups: total sleep time | Day 2
  total sleep time in hours and minutes
Comparison of sleep characterization between the two groups: number of sleep cycles | Day 2
  number of sleep cycles
Comparison of sleep characterization between the two groups: time spent awake during the night | Day 2
  time spent awake during the night
Comparison of sleep characterization between the two groups: index of micro-awakenings | Day 2
  index of micro-awakenings
Comparison of sleep characterization between the two groups: distribution of different sleep stages in time | Day 2
  distribution of different sleep stages in time
Comparison of sleep characterization between the two groups: distribution of different sleep stages in percentage | Day 2
  distribution of different sleep stages in percentage
Comparison of sleep characterization between the two groups: index of periodic movements | Day 2
  the index of periodic movements
Comparison of sleep characterization between the two groups: index of hypopnea | Day 2
  index of hypopnea (central and obstructive components)
Comparison of memory scores at the overnight retention test between the two groups | Day 2
  The memory scores are combined to compute a total score
symptoms of an underlying epileptic syndrome | Month 5
  The score on the questionnaire aiming at discovering potential symptoms of an underlying epileptic syndrome
sleep spindles in different sleep stages | day 2
  The number and the density of sleep spindles in different sleep stages
results of the cognitive reserve inventory (CRIq) | month 5
  Correlation between the frequency of epileptiform activity, the score on the epilepsy questionnaire and the index of micro-awakenings in the different sleep stages and: the results of the cognitive reserve inventory (CRIq)
speed of cognitive decline. | month 5
  Correlation between the frequency of epileptiform activity, the score on the epilepsy questionnaire and the index of micro-awakenings in the different sleep stages and: the speed of cognitive decline.
density of sleep spindles in the different sleep stages | month 5
  Correlation between the frequency of epileptiform activity, the score on the epilepsy questionnaire and the index of micro-awakenings in the different sleep stages and: the density of sleep spindles in the different sleep stages

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Dahan, PHD, Study Director — Centre de Recherches sur la Cognition Animale (CRCA), UMR CNRS 5169
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France